CLINICAL TRIAL: NCT07018739
Title: Efficacy of Using Mesenchymal Stem Cells With Therapeutic Hypothermia in Infants With Perinatal Hypoxic-Ischemic Encephalopathy: A Double Blind, Randomized Controlled Trial
Brief Title: Mesenchymal Stem Cells With Cooling Therapy for Infants With Hypoxic-Ischemic Encephalopathy
Acronym: SiSTEM-NEO
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 213/2025
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hypoxic-Ischemic Encephalopathy, Neonatal; Brain Injuries, Hypoxic-Ischemic
Keywords: Perinatal HIE; Mesenchymal stem cells; Wharton's jelly; therapeutic hypothermia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Injuries | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational product (MSCs or placebo) prepared by laboratory staff not involved in care or assessments. Syringes are identical in appearance and labeled only with subject codes. Clinical staff, investigators, and assessors remain blinded. Emergency unblinding allowed if medically necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wharton's jelly-derived mesenchymal stem cells (Experimental): A total of three IV infusions of MSCs will be administered, one dose per day for three consecutive days, starting within the first 10 days of life, following the completion of TH.
  Interventions: Biological: Wharton's jelly-derived mesenchymal stem cells
- Placebo (Placebo Comparator): A total of three IV infusions of 0.9%NSS will be administered, one dose per day for three consecutive days, starting within the first 10 days of life, following the completion of TH.
  Interventions: Drug: 0.9 % Normal Saline

INTERVENTIONS:
Biological: Wharton's jelly-derived mesenchymal stem cells — MSCs (2x10^6 cells/kg) in 10 mL 0.9%normal saline administered intravenously within 10 days, postnatally after TH completion, every 24 hours for 3 consecutive days
  Other Names: mesenchymal stem cells
  Arms: Wharton's jelly-derived mesenchymal stem cells
Drug: 0.9 % Normal Saline — 0.9% normal saline 10 mL administered intravenously within 10 days, postnatally after TH completion, every 24 hours for 3 consecutive days
  Other Names: 0.9%NSS
  Arms: Placebo

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE) is a serious condition in newborns caused by lack of oxygen and blood flow around the time of birth. Standard treatment with cooling therapy (therapeutic hypothermia) lowers the risk of death or disability, but many infants still suffer long-term problems.

This study will test whether adding stem cell therapy after cooling can further improve outcomes. The stem cells are taken from donated human placentas (Wharton's jelly-derived mesenchymal stem cells, MSCs). The cells are prepared under strict laboratory standards and checked for safety.

Infants with moderate to severe HIE who have completed cooling will be randomly assigned to receive either three intravenous infusions of MSCs or placebo within the first 10 days of life. Each infusion is given over about 30 minutes while the infant is closely monitored.

Researchers will follow participants for up to 2 years. The main outcome is whether MSC treatment can reduce the combined risk of death or serious developmental delay at 1 year of age. The study will also track brain MRI findings, safety events, and developmental progress at 2 years.

DETAILED DESCRIPTION:
Perinatal hypoxic-ischemic encephalopathy (HIE) is a major cause of neonatal death and long-term disability worldwide. Therapeutic hypothermia (TH) is the established standard of care for term and near-term infants with moderate to severe HIE. Large randomized trials and systematic reviews have demonstrated that TH significantly reduces the combined outcome of death or major neurodevelopmental disability at 18 months of age (relative risk 0.75; 95% confidence interval 0.68-0.83). However, despite this benefit, many infants continue to have poor outcomes. Importantly, a recent meta-analysis indicated that in upper-middle-income countries, the effect of TH was smaller and did not reach statistical significance (RR 0.67; 95% confidence interval 0.41-1.09), underscoring the need for effective adjunctive treatments.

Mesenchymal stem cells (MSCs) derived from Wharton's jelly of the human umbilical cord have emerged as a promising adjunctive therapy. Preclinical studies demonstrate that MSCs exert neuroprotective and regenerative effects via anti-inflammatory, anti-apoptotic, and trophic mechanisms. Early-phase clinical studies of cord blood or MSC products in neonatal HIE have shown feasibility and acceptable safety, with signals suggesting improved neurological recovery. Nevertheless, controlled trials specifically testing MSCs after completion of TH in neonates are lacking.

This study is a pilot, randomized, double-blind, placebo-controlled trial to evaluate the feasibility, safety, and potential efficacy of repeated intravenous infusions of Wharton's jelly-derived allogeneic MSCs in neonates with moderate to severe perinatal HIE who have completed TH. Forty infants (gestational age ≥34 weeks, postnatal age ≤10 days) will be randomized in a 1:1 ratio to receive either MSCs or placebo.

The intervention group will receive three intravenous doses of MSCs (2 × 10^6 cells/kg per dose, suspended in normal saline) administered over approximately 30 minutes. The control group will receive equivalent volumes of placebo (normal saline). Infants, parents, and treating clinicians will remain blinded to allocation.

All cell products are prepared in a GMP-compliant cleanroom facility with rigorous quality control testing, including sterility, endotoxin, mycoplasma, viability, morphology, immunophenotype, and karyotype. Donor placental tissue undergoes standard infectious disease screening.

Participants will be continuously monitored during and after infusion in the neonatal intensive care unit. Prespecified safety endpoints include fever, sepsis, hemodynamic instability, seizure control, acute liver failure, acute kidney injury, thrombosis, and death. A Data Safety Monitoring Board (DSMB) will review interim safety data at 25%, 50%, and 75% enrollment, and at 50% of 1-year follow-up. Predefined stopping rules will apply if significant safety concerns are identified.

The primary outcome is the composite of death or neurodevelopmental disability at 1 year of age, defined by Bayley Scales of Infant and Toddler Development, Fourth Edition (BSID-IV) cognitive, language, or motor scores <70. Secondary outcomes include hospital outcomes, brain MRI at 1 month (scored by Weeke criteria), HLA antibody formation at 9-12 months, and neurodevelopmental status at 2 years.

This pilot trial is designed to establish feasibility, evaluate safety, and generate preliminary efficacy estimates to inform future multicenter trials. All infants will receive standard TH and follow-up care, with the investigational therapy given only after cooling to test whether MSCs can further reduce death or disability in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Term and late-preterm infants (gestational age ≥34 weeks)
* Diagnosed with moderate to severe HIE based on modified Sarnat staging
* Received TH per standard protocol
* Parental consent obtained

Exclusion Criteria:

* Major congenital anomalies or genetic syndromes
* Severe sepsis or active infection
* Severe coagulopathy or bleeding disorders
* Multi-organ failure

Ages: 4 Days to 9 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Death or neurological disability | At 12 months of age
  Including any causes of deaths. Neurological disability is defined by Bayley Scales of Infant Development-IV <70 (ranging from 40 to 160, with higher scores indicating better neurodevelopmental outcomes)

SECONDARY OUTCOMES:
Death or neurological disability | At 24 months postnatal age
  Any causes of death. Neurological disability is defined as Bayley Scales of Infant Development-IV <70 (ranging from 40 to 160, with higher scores indicating better neurodevelopmental outcomes)
MR-detected brain injury | At 1 month of age
  Brain injury detected by Weeke MRI score on brain MRI (total score range 0-57; higher scores indicate worse outcomes).
Severe adverse events | From first study infusion until hospital discharge, up to 12 months
  One of these adverse events occurring after drug initiation:
  Hemodynamic instability (persistent HR >180 beats per minute, BP <5th %tile for gestational age and postnatal age, require new treatment (volume resuscitation/inotropic agents/vasopressor agents) Acute liver failure (new-onset of hyperbilirubinemia with INR ≥3 with no response to vitamin K administration) Thrombosis (any events such as renal vein thrombosis, stroke) Death before discharge
HLA antibody formation | At 9-12 months of age
  Presence of anti-HLA antibodies assessed by panel-reactive antibody (PRA) testing.
Length of birth hospitalization | Through hospital discharge, up to 12 months
  Total days from birth to hospital discharge.
Incidence of infection | Through hospital discharge, up to 12 months
  Culture-proven infection requiring antimicrobial therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ratchada Kitsommart, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying published results (e.g., baseline demographics, adverse events, primary and secondary outcomes including Bayley-IV scores and Weeke MRI scores).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the primary results, available for 5 years
Access Criteria: Data will be available upon reasonable request to the Principal Investigator at Siriraj Hospital, subject to institutional review and data-sharing agreements.

REFERENCES:
- [Background] Xu J, Feng Z, Wang X, Xiong Y, Wang L, Ye L, Zhang H. hUC-MSCs Exert a Neuroprotective Effect via Anti-apoptotic Mechanisms in a Neonatal HIE Rat Model. Cell Transplant. 2019 Dec;28(12):1552-1559. doi: 10.1177/0963689719874769. Epub 2019 Sep 12. PMID 31512502
- [Result] Bruschettini M, Romantsik O, Moreira A, Ley D, Thebaud B. Stem cell-based interventions for the prevention of morbidity and mortality following hypoxic-ischaemic encephalopathy in newborn infants. Cochrane Database Syst Rev. 2020 Aug 19;8(8):CD013202. doi: 10.1002/14651858.CD013202.pub2. PMID 32813884
- [Result] Teo EJ, Jones LE, Wixey JA, Boyd RN, Colditz PB, Bjorkman ST. Combined hypothermia and mesenchymal stem cells in animal models of neonatal hypoxic-ischaemic encephalopathy: a systematic review. Pediatr Res. 2022 Jul;92(1):25-31. doi: 10.1038/s41390-021-01716-y. Epub 2021 Sep 4. PMID 34482377
- [Result] Ahn SY, Chang YS, Sung DK, Sung SI, Park WS. Hypothermia broadens the therapeutic time window of mesenchymal stem cell transplantation for severe neonatal hypoxic ischemic encephalopathy. Sci Rep. 2018 May 16;8(1):7665. doi: 10.1038/s41598-018-25902-x. PMID 29769612
- [Result] Terada K, Sasaki M, Nagahama H, Kataoka-Sasaki Y, Oka S, Ukai R, Yokoyama T, Iizuka Y, Sakai T, Fukumura S, Tsugawa T, Kocsis JD, Honmou O. Therapeutic efficacy of intravenous infusion of mesenchymal stem cells in rat perinatal brain injury. Pediatr Res. 2023 Dec;94(6):1921-1928. doi: 10.1038/s41390-023-02717-9. Epub 2023 Jul 8. PMID 37422495
- [Result] van Velthoven CT, Kavelaars A, van Bel F, Heijnen CJ. Mesenchymal stem cell treatment after neonatal hypoxic-ischemic brain injury improves behavioral outcome and induces neuronal and oligodendrocyte regeneration. Brain Behav Immun. 2010 Mar;24(3):387-93. doi: 10.1016/j.bbi.2009.10.017. Epub 2009 Oct 31. PMID 19883750
- [Result] van Velthoven CT, Kavelaars A, van Bel F, Heijnen CJ. Repeated mesenchymal stem cell treatment after neonatal hypoxia-ischemia has distinct effects on formation and maturation of new neurons and oligodendrocytes leading to restoration of damage, corticospinal motor tract activity, and sensorimotor function. J Neurosci. 2010 Jul 14;30(28):9603-11. doi: 10.1523/JNEUROSCI.1835-10.2010. PMID 20631189
- [Result] Wagenaar N, de Theije CGM, de Vries LS, Groenendaal F, Benders MJNL, Nijboer CHA. Promoting neuroregeneration after perinatal arterial ischemic stroke: neurotrophic factors and mesenchymal stem cells. Pediatr Res. 2018 Jan;83(1-2):372-384. doi: 10.1038/pr.2017.243. Epub 2017 Nov 1. PMID 28949952
- [Result] Ahn SY, Chang YS, Sung DK, Sung SI, Ahn JY, Park WS. Pivotal Role of Brain-Derived Neurotrophic Factor Secreted by Mesenchymal Stem Cells in Severe Intraventricular Hemorrhage in Newborn Rats. Cell Transplant. 2017 Jan 24;26(1):145-156. doi: 10.3727/096368916X692861. Epub 2016 Aug 16. PMID 27535166
- [Result] Lalu MM, McIntyre L, Pugliese C, Fergusson D, Winston BW, Marshall JC, Granton J, Stewart DJ; Canadian Critical Care Trials Group. Safety of cell therapy with mesenchymal stromal cells (SafeCell): a systematic review and meta-analysis of clinical trials. PLoS One. 2012;7(10):e47559. doi: 10.1371/journal.pone.0047559. Epub 2012 Oct 25. PMID 23133515
- [Result] Mintoft A, Vallatos A, Robertson NJ. Mesenchymal Stromal Cell therapy for Hypoxic Ischemic Encephalopathy: Future directions for combination therapy with hypothermia and/or melatonin. Semin Perinatol. 2024 Aug;48(5):151929. doi: 10.1016/j.semperi.2024.151929. Epub 2024 Jun 13. PMID 38902120
- [Result] Dezawa M, Kanno H, Hoshino M, Cho H, Matsumoto N, Itokazu Y, Tajima N, Yamada H, Sawada H, Ishikawa H, Mimura T, Kitada M, Suzuki Y, Ide C. Specific induction of neuronal cells from bone marrow stromal cells and application for autologous transplantation. J Clin Invest. 2004 Jun;113(12):1701-10. doi: 10.1172/JCI20935. PMID 15199405
- [Result] Uccelli A, Moretta L, Pistoia V. Mesenchymal stem cells in health and disease. Nat Rev Immunol. 2008 Sep;8(9):726-36. doi: 10.1038/nri2395. PMID 19172693
- [Result] Braccioli L, Heijnen CJ, Coffer PJ, Nijboer CH. Delayed administration of neural stem cells after hypoxia-ischemia reduces sensorimotor deficits, cerebral lesion size, and neuroinflammation in neonatal mice. Pediatr Res. 2017 Jan;81(1-1):127-135. doi: 10.1038/pr.2016.172. Epub 2016 Sep 15. PMID 27632779
- [Result] Kaminski N, Koster C, Mouloud Y, Borger V, Felderhoff-Muser U, Bendix I, Giebel B, Herz J. Mesenchymal Stromal Cell-Derived Extracellular Vesicles Reduce Neuroinflammation, Promote Neural Cell Proliferation and Improve Oligodendrocyte Maturation in Neonatal Hypoxic-Ischemic Brain Injury. Front Cell Neurosci. 2020 Dec 10;14:601176. doi: 10.3389/fncel.2020.601176. eCollection 2020. PMID 33362471
- [Result] Nabetani M, Shintaku H, Hamazaki T. Future perspectives of cell therapy for neonatal hypoxic-ischemic encephalopathy. Pediatr Res. 2018 Jan;83(1-2):356-363. doi: 10.1038/pr.2017.260. Epub 2017 Nov 8. PMID 29016557